CLINICAL TRIAL: NCT01145664
Title: A Multi-Center Clinical Trial To Evaluate Chinese Herbal Medicines in the Treatment of Severe Hand-foot-mouth Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing YouAn Hospital (Other)
Collaborators: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government); China Academy of Chinese Medical Sciences (Other); Beijing University of Chinese Medicine (Other)
Responsible Party: Xiuhui Li, Beijing YouAn Hospital，Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200907001-3; NCT01314794 (obsolete NCT alias)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-05

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Chinese medicines; Severe hand-foot-mouth diseases; effectiveness; safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — reduning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Western therapy (Active Comparator)
  Interventions: Drug: Western therapy
- Herbal concentrate-granules plus western therapy (Experimental)
  Interventions: Drug: Herbal concentrate-granules plus western therapy
- Reduning Injection plus western therapy (Experimental)
  Interventions: Drug: Reduning Injection plus western therapy

INTERVENTIONS:
Drug: Herbal concentrate-granules plus western therapy — Intervention time: 7-10 days; Follow-up time: 5 days.
  Arms: Herbal concentrate-granules plus western therapy
Drug: Reduning Injection plus western therapy — Intervention time: 7-10 days; Follow-up time: 5 days.
  Arms: Reduning Injection plus western therapy
Drug: Western therapy — Intervention time: 7-10 days; Follow-up time: 5 days.
  Arms: Western therapy

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Chinese herbal medicines for severe hand-foot-mouth disease.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of severe hand-foot-mouth disease patients according to hand-foot-mouth disease treatment guidelines 2010 issued by China's Ministry of Health
2. not more than 24 hours of occurrence of severe symptoms
3. age of 1-13 years
4. Patients or their guardians agree to participate in this study and signed the informed consent form

Exclusion Criteria:

1. Suffering from neurogenic pulmonary edema, heart or lung failure.
2. Complicated with other serious diseases such as chronic hepatitis, congenital heart disease, acute or chronic nephritis and blood diseases, etc
3. the history of allergies on Chinese medicine
4. the history of mild increase of blood bilirubin hemolysis (or uric bravery former positive) phenomenon
5. using hormonal therapy
6. Attending other clinical studies on hand-foot-mouth disease
7. Patients or their guardians suffering from mental illness

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 390 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
incidence of complications | 15 days
incidence of critically ill patients | 15 days

SECONDARY OUTCOMES:
case fatality rate | 15 days
time of symptom disappearance | 15 days
time of bringing down a fever | 15 days
length of stay | 15 days
dose and usage of hormones | 15 days
safety outcome(adverse effects) | 15 days

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Guangzhou Women and Children Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Kaifeng Municipal Children's Hospital, Kaifeng, Henan
  - Hunan Provincial Children's Hospital, Changsha, Hunan
  - Anhui Provincial Children's Hospital, Anhui
  - Beijing YouAn Hospital，Capital Medical University, Beijing

REFERENCES:
- [Derived] Li XH, Li SJ, Xu Y, Wei D, Shi QS, Zhu QX, Yang T, Ding JB, Tian YM, Huang JH, Wang K, Wen T, Zhang X. Effect of integrated Chinese and Western medicine therapy on severe hand, foot and mouth disease: A prospective, randomized, controlled trial. Chin J Integr Med. 2017 Dec;23(12):887-892. doi: 10.1007/s11655-016-2504-3. Epub 2016 Jul 9. PMID 27392481